CLINICAL TRIAL: NCT02552069
Title: The Verification Study on the Early Fixation/ Stability of Tritanium Cup
Brief Title: Tritanium® Study in Japan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stryker Japan K.K. (Industry)
Responsible Party: Sponsor
Other Study IDs: SJCR-OR-1505
Record Dates: First submitted 2015-08-10; First posted 2015-09-16 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Avascular Necrosis of the Femoral Head
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Femur Head Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tritanium® cup
  Interventions: Device: Tritanium® cup

INTERVENTIONS:
Device: Tritanium® cup

SUMMARY:
The purpose of this study is to evaluate early fixation and stability of the Tritanium cup. It is expected that the Tritanium® cup will be equal to or better than conventional cementless cups in early fixation/stability and meet the expectations of Japanese surgeons.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a candidate for a primary Total Hip Arthroplasty (THA).
2. Patient who has diagnosis of secondary osteoarthritis, avascular necrosis and rheumatoid arthritis.
3. Patient whose age is 20 or over.
4. Patient who signed an Institutional Review Board (IRB)-approved, study specific Informed Patient Consent Form.
5. Patient who is willing and able to comply with postoperative scheduled evaluations.

Exclusion Criteria:

1. Patient who has a bacterial infectious disease or has a high risk of a bacterial infection.
2. Patient who requires revision surgery of a previously implanted total hip arthroplasty.
3. Patient who is morbidly obese, defined as having a Body Mass Index (BMI) > 40.
4. Patient who is or may be pregnant female.
5. Patient who has neuromuscular or neurosensory deficiency, which limits ability to evaluate the safety and efficacy of the device.
6. Patient with diagnosed systemic disease (i.e. Paget's disease, renal osteodystrophy), which limits ability to evaluate the safety and efficacy of the device.
7. Patient who is immunologically suppressed or receiving chronic steroids, which limits ability to evaluate the safety and efficacy of the device.
8. Patients who is judged ineligible with specific reason by primary doctor.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who has diagnosis of secondary osteoarthritis, avascular necrosis and rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in implantation position(angle) of the cup | Baseline, intraoperative, 3 months, 6 months and 12 months

SECONDARY OUTCOMES:
Change in Japanese Orthopaedic Association (JOA) score | Baseline, 3 months, 6months and 12 months
Change in Quality of Life as assessed by Euro QOL 5 Dimension (EQ-5D) | Pre-operation, 3 months, 6months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yasuyuki Inatsugu, Study Director — Stryker Japan
Locations (1):
- RINKU General Medical Center, Izumisano, Osaka, Japan